CLINICAL TRIAL: NCT02819674
Title: The Chinese Early-onset Hypertension Study (CHESS)
Acronym: CHESS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Lei.Song@NCCD, MD, ph.D, China National Center for Cardiovascular Diseases
Other Study IDs: CEHS-2016
Record Dates: First submitted 2016-05-20; First posted 2016-06-30 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Hypertension
Keywords: hypertension; early onset; target organ damage
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples are collected after 12-hour overnight fast and biological variables are determined. Genomic DNA is isolated from leukocytes according to a standard procedure.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- early-onset hypertension: early-onset hypertension patients recruited in Chinese multiple centers

SUMMARY:
Hypertension (HTN) is the most important cardiovascular risk factor which is responsible for 50% of cardiovascular morbidity and mortality, and also a substantial public health problem affecting approximately 1/4 of the adult population in industrialized societies and over 1 billion people worldwide. Chronically elevated blood pressure without well control puts people at increased risk of target organ damages, including stroke, myocardial infarction, congestive heart failure, end-stage renal disease, blindness, and death. Especially, these damages are dramatically more severe in the early-onset hypertensive population.

DETAILED DESCRIPTION:
In this study, the hypertensive individuals are consecutively recruited from multiple centers, with an early onset age (less than 40 when diagnosed). A complete clinical history (information on history of hypertension, demographic characteristics, personal and family medical history) are collected by a trained staff using a standardized questionnaire on the first day of baseline observation, and physical examination are also collected in a standard procedure. Blood samples are collected after 12-hour overnight fast and biological variables are determined. Genomic DNA is isolated from leukocytes according to a standard procedure. The individuals will receive follow-up in an ordinal system. The investigators will focus on the clinical and genetic features, genotype-phenotype correlations and influencing factors of prognosis in Chinese early-onset hypertension patients.

ELIGIBILITY:
Inclusion Criteria:

* In accordance with the diagnosis of hypertension (BP≥140/90mmHg), and less than 40 years when diagnosed

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Between October 2012 and December 2020(anticipated) recruited from multiple centers in China, in accordance with the diagnosis of hypertension, and less than 40 years when diagnosed
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2012-10; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
primary mortality of early-onset hypertension | through study completion, an average of 5 years
  the primary mortality of early-onset hypertension

SECONDARY OUTCOMES:
secondary outcomes of heart | through study completion, an average of 5 years
  The incidence rate of left ventricular hypertrophy, myocardial infarction, congestive heart failure, and arrhythmia.
secondary outcomes of brain | through study completion, an average of 5 years
  The incidence rate of stroke (include cerebral hemorrhage and cerebral ischemia)
secondary outcomes of kidney | through study completion, an average of 5 years
  The incidence rate of hypertensive renal injure and end-stage renal disease
secondary outcomes of eyes | through study completion, an average of 5 years
  The incidence rate of hypertensive eye injure

CONTACTS AND LOCATIONS:
Overall Officials: Lei Song, MD.& PhD., Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided